CLINICAL TRIAL: NCT00639613
Title: Exspression of Prohormone Convertase 1 and 2 in Small Intestinal Endocrine Mucosa Cells in Patients With Type 2 Diabetes
Brief Title: The Role of Small Intestinal Endocrine Cells in Type 2 Diabetic Hyperglucagonemia
Acronym: T2DM-PC1-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Head of Diabetes Research Division, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-B-2007-031
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with type 2 diabetes
  Interventions: Procedure: Double-balloon enteroscopy; Other: Standard meal test
- 2: Healthy subjects
  Interventions: Procedure: Double-balloon enteroscopy; Other: Standard meal test

INTERVENTIONS:
Procedure: Double-balloon enteroscopy — Double-balloon enteroscopy allows for the entire gastrointestinal tract to be visualized in real time. The technique involves the use of a balloon at the end of a special enteroscope camera and an overtube, which is also fitted with a balloon. The procedure is usually done with the use of conscious sedation. The enteroscope and overtube are inserted through the mouth and passed in conventional fashion (that is, as with gastroscopy) into the small bowel. Following this, the endoscope is advanced a small distance in front of the overtube and the balloon at the end is inflated. Using the assistance of friction at the interface of the enteroscope and intestinal wall, the small bowel is accordioned back to the overtube. The overtube balloon is then deployed, and the enteroscope balloon is deflated. The process is then continued until the entire small bowel is visualized. Double-balloon enteroscopy allows for the sampling or biopsying of small bowel mucosa.
Other: Standard meal test — Liquid meal consisting of 100 g "Ny NAN" dissolved in 300 ml water (ca. 5000 kJ) to be ingested over 5 minutes. Blood will be sampled for 4 hours following ingestion. Samples are centrifuges and plasma will be analysed for glucagon, GLP-1, GIP, insulin and C-peptide concentrations.

SUMMARY:
The purpose of this study is to determine whether excessive secretion of glucagon in type 2 diabetes originates from the pancreatic alpha-cells or endocrine cells in the mucosa of the small intestinal.

DETAILED DESCRIPTION:
Hyperglucagonemia contributes significantly to the hyperglycemia characterizing patients with Type 2 diabetes. Fasting hyperglucagonemia induces hepatic glucose release resulting in elevated fasting levels of plasma glucose. Furthermore, lack of postprandial suppression of glucagon secretion - exchanged for a paradoxical postprandial hypersecretion of glucagon - results in increased levels of postprandial plasma glucose. Additionally, type 2 diabetes is characterized by decreased postprandial responses of the insulinotropic (and glucagonostatic) peptide hormone glucagon-like peptide-1 (GLP-1). Recent studies from our group suggest that the intestines are involved in the diminshed suppression of glucagon following ingestion of nutrients. Thus, suppression of glucagon during oral glucose ingestion diminishes and reverses to stimulation while suppression during intravenous administered glucose sustains along with development of glucose intolerance. In the small intestines mucosal endocrine L-cells secrete GLP-1, which is processed from its precursor, proglucagon, by prohormone convertase 1 (PC1). In the pancreatic alpha-cells proglucagon is processed to glucagon via prohormone convertase 2 (PC2). We plan to examine biopsies from the mucosa of the small intestines from patients with type 2 diabetes and from healthy subjects for glucagon production. Furthermore, the volunteers will be subjected to a standard meal test in order to correlate the gene expression studies with the level of postprandial hyperglucagonemia of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 3 months
* Normal hemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT/ASAT > 2 x normal range)
* Diabetic nephropathy (se-creatinin > 130 µM and/or albuminuriu)
* Treatment with medication that can not be stopped for12 hours

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- Department of Internal Medicine F' laboratory, Hellerup, Copenhagen County, Denmark